CLINICAL TRIAL: NCT06128564
Title: A Two-Part, Open-Label Systemic Gene Delivery Study to Evaluate the Safety and Expression of RO7494222 (SRP-9001) in Subjects Under the Age of Four With Duchenne Muscular Dystrophy
Brief Title: A Gene Delivery Study to Evaluate the Safety and Expression of Delandistrogene Moxeparvovec in Participants Under the Age of Four With Duchenne Muscular Dystrophy (DMD)
Acronym: ENVOL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BN43881; 2022-000691-19 (EudraCT Number); 2023-509901-57-00 (EU CTIS Number)
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: DMD; Duchenne; Dystrophin; Gene-Delivery; Pediatric
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Delandistrogene Moxeparvovec (Experimental): Participants will receive a single intravenous (IV) infusion of delandistrogene moxeparvovec on Day 1.
  Interventions: Genetic: delandistrogene moxeparvovec

INTERVENTIONS:
Genetic: delandistrogene moxeparvovec — Single IV infusion of delandistrogene moxeparvovec
  Other Names: SRP-9001; ELEVIDYS; RO7494222; delandistrogene moxeparvovec-rokl

SUMMARY:
This open-label, single-arm study will evaluate the safety and expression of delandistrogene moxeparvovec in participants with DMD. Participants will be in the study for approximately 264 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Cohort A: >=3 years of age to <4 years of age
* Cohort B: >=2 years of age to <3 years of age
* Has a definitive diagnosis of DMD prior to screening based on documentation of clinical findings and prior confirmatory genetic testing using a clinical diagnostic genetic test
* Able to cooperate with age-appropriate motor assessment testing
* A pathogenic frameshift mutation or premature stop codon contained between exons 18 and 79 (inclusive)

Exclusion Criteria:

* Exposure to gene therapy, investigational medication, or any treatment designed to increase dystrophin expression, within protocol-specified time limits
* Recombinant Adeno-Associated Virus Serotype rh74 (rAArh74) antibody titers are elevated, as per protocol-specified criteria
* Receiving regular oral corticosteroids as a treatment for DMD or planning to receive oral corticosteroids as a treatment for DMD within 1 year of baseline
* Presence of any other clinically significant illness, medical condition, or requirement for chronic drug treatment that in the opinion of the Investigator creates unnecessary risk for gene transfer
* Medical condition or extenuating circumstance that, in the opinion of the investigator, might compromise the participant's ability to comply with the protocol required testing or procedures, or compromise the participant's well-being or safety, or clinical interpretability

Other inclusion or exclusion criteria could apply

Ages: 2 Years to 3 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2030-02-28 (Estimated); Study Completion 2034-01-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with a Treatment-emergent Adverse Event (TEAE), Serious Adverse Event (SAE), and Adverse Event of Special Interest (AESI) | Baseline up to Week 260

SECONDARY OUTCOMES:
Change in Quantity of Delandistrogene Moxeparvovec Dystrophin as Measured by Western Blot | Baseline, Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- Chr de La Citadelle, Liège, Belgium
- Hôpital Necker-Enfants Malades, Paris, France
- Universitätsklinikum Essen, Essen, Germany
- PU A. Gemelli, Università Cattolica del Sacro Cuore, Rome, Lazio, Italy
- Hospital Sant Joan De Deu, Esplugues de Llobregas, Barcelona, Spain
- United Kingdom (2):
  - Great Ormond Street Hospital for Children, London
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing